CLINICAL TRIAL: NCT01776697
Title: A Randomized, Open-labeled, Comparative 3-way Crossover Study to Compare the Pharmacokinetic Characteristics and Food Effect of Pelubiprofen (30mg) Tablet IR TID and Pelubiprofen SR (as a Pelubiprofen 90 mg) Tablet QD in Healthy Subjects
Brief Title: Phase 1 Study to Compare the Pharmacokinetic Characteristics and Food Effect of Pelubiprofen (30mg) Tablet IR TID and Pelubiprofen SR (as a Pelubiprofen 90 mg) Tablet QD in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: DW330SR-1001(Ver2.2)
Record Dates: First submitted 2013-01-22; First posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
MeSH Terms: interventions — pelubiprofen; Tablets

ARMS (3):
- pelubiprofen (30mg) tablet IR TID, fasting (Active Comparator)
  Interventions: Drug: pelubiprofen (30mg) tablet IR
- pelubiprofen (30mg) tablet IR TID, fed (Active Comparator)
  Interventions: Drug: pelubiprofen (30mg) tablet IR
- pelubiprofen SR (as a pelubiprofen 90 mg) tablet QD (Experimental)
  Interventions: Drug: pelubiprofen SR (as a pelubiprofen 90 mg) tablet

INTERVENTIONS:
Drug: pelubiprofen (30mg) tablet IR
  Arms: pelubiprofen (30mg) tablet IR TID, fasting; pelubiprofen (30mg) tablet IR TID, fed
Drug: pelubiprofen SR (as a pelubiprofen 90 mg) tablet
  Arms: pelubiprofen SR (as a pelubiprofen 90 mg) tablet QD

SUMMARY:
A randomized, open-labeled, comparative 3-way crossover study to compare the pharmacokinetic characteristics and food effect of pelubiprofen (30mg) tablet IR TID and pelubiprofen SR (as a pelubiprofen 90 mg) tablet QD in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Healthy males aged 20~45 years
2. weight over 45 kg, ideal body weight ±20%[Ideal weight] = [Height(cm)-100] X 0.9
3. Subjects who voluntarily agreed with written consent

Exclusion Criteria:

1. Patients with acute disorder within 28 days before clinical trial drugs administration
2. History of disorders(inflammatory GI tract disease, stomach ulcer, gastrectomy, liver disease) which can affect ADME of drugs
3. Patients with active GI tract, cardiovascular, respiratory, renal, endocrinal, haematological, central nerval, psychiatric disease or malignant tumor

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
AUC of pelubiprofen(30mg) tablet IR TID | 0, 1, 2, 8, 9, 15, 16, 22 day
AUC of pelubiprofen SR (as a pelubiprofen 90 mg) tablet QD | 0, 1, 2, 8, 9, 15, 16, 22 day
Cmax of pelubiprofen(30mg) tablet IR TID | 0, 1, 2, 8, 9, 15, 16, 22 day
Cmax of pelubiprofen SR (as a pelubiprofen 90 mg) tablet QD | 0, 1, 2, 8, 9, 15, 16, 22 day